CLINICAL TRIAL: NCT06916065
Title: A Phase 1, Open-Label, Single and Multiple Dose Study to Investigate the Safety, Tolerability, and Relative Bioavailability of Single and Multiple Weekly Subcutaneous Doses of Eloralintide, and Single and Multiple Weekly Subcutaneous Doses of Eloralintide With Tirzepatide in Participants With Overweight or Obesity
Brief Title: A Study of Eloralintide (LY3841136) and Eloralintide With Tirzepatide in Participants With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27353; J3R-MC-YDAE (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eloralintide and Tirzepatide-Cohorts A-D (Experimental): Eloralintide and Tirzepatide administered subcutaneously (SC)
  Interventions: Drug: Eloralintide and Tirzepatide
- Eloralintide-Cohorts E and F (Experimental): Eloralintide administered SC
  Interventions: Drug: Eloralintide

INTERVENTIONS:
Drug: Eloralintide and Tirzepatide — Administered SC
  Other Names: LY3841136
  Arms: Eloralintide and Tirzepatide-Cohorts A-D
Drug: Eloralintide — Administered SC
  Other Names: LY3841136
  Arms: Eloralintide-Cohorts E and F

SUMMARY:
The purpose of this study is to evaluate how well eloralintide and eloralintide with tirzepatide is tolerated and what side effects may occur in participants with overweight or obesity. The study drug will be administered subcutaneously (SC) (under the skin). Blood tests will be performed to check how much eloralintide and eloralintide with tirzepatide get into the bloodstream and how long it takes the body to eliminate it.

There will be 6 cohorts. The study will last up to approximately 26 weeks, excluding screening for Cohorts A and B, 11 weeks for Cohorts C and D, and 12 weeks for Cohorts E and F.

ELIGIBILITY:
Inclusion Criteria:

* Have safety laboratory test results within normal reference range for the population or investigative site, or results with acceptable deviations that are judged to be not clinically significant by the investigator. Participants with a history of thyroid disease or on thyroid medication will need to be biochemically euthyroid as assessed by measuring thyroid stimulating hormone at screening
* Have a body mass index (BMI) within the range of 27.0 to 40.0 kilogram per square meter (kg/m²), inclusive
* Have had a stable weight for the 3 months prior to screening, that is, less than 5% body weight change

Exclusion Criteria:

* Have known allergies to related compounds of eloralintide or tirzepatide, or any of the components of the formulations
* Have significant previous or current history of comorbidities capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data
* Have been diagnosed with Type 1 or Type 2 diabetes mellitus, or have glycated hemoglobin greater than or equal to 6.5% or 48 millimole per mole (mmol/mol)
* Have a history of any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Have a history or presence of a gastrointestinal (GI) disorder or previous surgery that impacts gastric emptying for example, gastric bypass surgery or pyloric stenosis
* Have obesity induced by other endocrinologic disorders for example, Cushing syndrome, or diagnosed monogenetic or syndromic forms of obesity for example, Melanocortin 4 Receptor deficiency or Prader Willi syndrome
* Have a history of hypocalcemia or hypercalcemia, or abnormal laboratory values for calcium or serum phosphorus
* Have a medical history or current evidence of clinically significant cardiac condition, as per the investigator, including:

  * second or third degree heart block
  * sick sinus syndrome
  * peripheral arterial circulatory disorders
  * valvular disease
  * cardiomyopathy, or
  * other clinically significant cardiac condition
* Have taken approved or investigational medication for weight loss, including GLP-1 RAs, within the previous 3 months of study screening
* Intend to use any weight loss medications during study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-01-19 (Actual); Study Completion 2026-01-19 (Actual)

PRIMARY OUTCOMES:
Cohorts A and B: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of Eloralintide and Tirzepatide | Day 106 Predose to Approximately Week 26
  PK: AUC of Eloralintide and Tirzepatide
Cohorts A and B: PK: Maximum Concentration (Cmax) of Eloralintide and Tirzepatide | Day 106 Predose to Approximately Week 26
  PK: Cmax of Eloralintide and Tirzepatide
Cohorts C and D: PK: AUC of Eloralintide and Tirzepatide | Baseline Up to Approximately Week 11
  PK: AUC of Eloralintide and Tirzepatide
Cohorts C and D: PK: Cmax of Eloralintide and Tirzepatide | Baseline Up to Approximately Week 11
  PK: Cmax of Eloralintide and Tirzepatide
Cohorts E and F: PK: AUC of Eloralintide | Day 8 Predose Up to Approximately Week 12
  PK: AUC of Eloralintide
Cohorts E and F: PK: Cmax of Eloralintide | Day 8 Predose Up to Approximately Week 12
  PK: Cmax of Eloralintide
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline Up to Approximately Week 26
  A summary of TEAEs and SAEs regardless of causality, will be reported in the Reported Adverse Events module

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Fortrea Clinical Research Unit, Daytona Beach, Florida
  - Fortrea Clinical Research Unit, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://trials.lilly.com/en-US/trial/590708